CLINICAL TRIAL: NCT06705101
Title: GABAPENTIN ATTENUATES THE PRESSOR RESPONSE TO DIRECT LARYNGOSCOPY AND TRACHEAL INTUBATION
Brief Title: Gabapentin and Pressor Response to Intubation
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, SYEDA AEMAN ZUBAIR, DR, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0842-2022-LNH-ERC
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Elective Surgical Patients; Blood Pressure
Keywords: Gabapentin; Laryngoscopy; Hemodynamic Stability; Pressor Response
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gabapentin Group (Group G): Participants receiving Gabapentin 300 mg as a pre-treatment. (Experimental): Gabapentin Group (Group G): Participants receiving Gabapentin 300 mg as a pre-treatment.
  Interventions: Drug: Gabapentin Group (Group G): Patients will receive 300 mg of oral Gabapentin
- Placebo Group (Group P): Participants receiving a placebo as a pre-treatment. (Placebo Comparator): Placebo Group (Group P): Participants receiving a placebo as a pre-treatment.
  Interventions: Other: Placebo Oral Tablet

INTERVENTIONS:
Drug: Gabapentin Group (Group G): Patients will receive 300 mg of oral Gabapentin — In this study, the intervention involves administering 300 mg of oral gabapentin to patients in the intervention group two hours prior to surgery, aiming to assess its efficacy in attenuating the pressor response to laryngoscopy and tracheal intubation.
  Arms: Gabapentin Group (Group G): Participants receiving Gabapentin 300 mg as a pre-treatment.
Other: Placebo Oral Tablet — The placebo group will receive an identical capsule without active medication, administered two hours before surgery, to compare its effects with those of gabapentin on the pressor response to laryngoscopy and tracheal intubation.
  Arms: Placebo Group (Group P): Participants receiving a placebo as a pre-treatment.

SUMMARY:
This study evaluates the effectiveness of oral gabapentin in reducing the pressor response (increased MAP, HR, and BP) during laryngoscopic intubation. It is a prospective, double-blind randomized controlled trial involving 144 patients undergoing elective surgery. Gabapentin 300 mg or placebo will be administered preoperatively, with hemodynamic parameters monitored before and after intubation. The study aims to determine if gabapentin attenuates the sympathetic stress response compared to placebo.

DETAILED DESCRIPTION:
Laryngoscopic tracheal intubation often triggers a significant sympathetic response, causing increased heart rate, blood pressure, and other hemodynamic changes, which can pose risks for patients with underlying cardiovascular or cerebrovascular conditions. While various methods and drugs have been employed to mitigate this pressor response, gabapentin-a GABA analog with multimodal effects-has shown promise in reducing such hemodynamic stress. This study aims to evaluate the effectiveness of oral gabapentin as a pretreatment to attenuate the sympathetic response during intubation.

The objective of this study is to compare the effectiveness of gabapentin versus placebo in reducing stress responses, such as mean arterial pressure (MAP), heart rate (HR), and blood pressure (BP), during general anesthesia with endotracheal intubation.

Study Design is Prospective, double-blind, randomized controlled trial and will be conducted in Department of Anesthesia, Liaquat National Hospital.

during 8 months. 144 patients (72 per group), calculated based on prior MAP data, with patients randomized into Gabapentin (Group G) and Placebo (Group P) Patients aged 18-59 years, ASA I or II, undergoing elective surgeries will be included.

Exclusion Criteria is difficult intubation, ASA III or higher, obesity, or use of antihypertensive or sedative drugs.

Participants will receive either 300 mg oral gabapentin or placebo 2 hours before surgery. Standard monitoring and anesthesia protocols will be followed, with blood pressure and heart rate recorded at baseline, 2 minutes, and 5 minutes post-intubation. The primary outcome is MAP, while secondary outcomes include systolic/diastolic BP and HR. Intravenous metoprolol will be administered if required for pressor responses.

SPSS v25 will be used for statistical analysis, with independent t-tests for quantitative data and chi-square tests for categorical variables. A p-value <0.05 will be considered statistically significant.

Hypothesis:

Null: Gabapentin does not attenuate the pressor response. Alternative: Gabapentin attenuates the pressor response.

Rationale:

Gabapentin's potential to modulate sympathetic responses during intubation offers a novel, multimodal approach to anesthesia management. While international studies exist, no local studies have been conducted, making this research vital for assessing its efficacy in the local population.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II patients (American Society of Anesthesiologists Physical Status Classification).
* Age between 18 and 59 years.
* Scheduled for elective surgery under general anesthesia with endotracheal intubation.

Exclusion Criteria:

* Anticipated difficult intubation.
* ASA III or greater.
* Patients with hiatus hernia or gastro-esophageal reflux disease (GERD).
* Body weight more than 20% of ideal body weight.
* Patients on antihypertensive drugs, sedatives, hypnotics, or antidepressants.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-16 (Estimated)

PRIMARY OUTCOMES:
Mean Arterial Pressure (MAP) | 2 minutes, and 5 minutes after laryngoscopy and tracheal intubation
  The primary outcome is the change in MAP before intubation, 2 minutes, and 5 minutes after laryngoscopy and tracheal intubation. The focus is on whether Gabapentin maintains MAP within 20 mmHg of the patient's baseline reading.

IPD SHARING:
Plan to Share IPD: No